CLINICAL TRIAL: NCT05287308
Title: Adjuvant AC Followed by Albumin-bound Paclitaxel Versus AC Followed by Taxanes in Breast Cancer: a Prospective, Multi-center, Real-world Study
Brief Title: Adjuvant Albumin-bound Paclitaxel Versus Taxanes in Breast Cancer: a Real-world Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Binghe Xu, Academician，Director of Department of Clinical Trial Center, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LQ009
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Epirubicin; pirarubicin; Cyclophosphamide; Albumin-Bound Paclitaxel; Paclitaxel; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AC followed by albumin-bound paclitaxel (Experimental): A (doxorubicin, epirubicin or pirarubicin) and C (cyclophosphamide) for 4 cycles followed by albumin-bound paclitaxel for 4 cycles.
  Interventions: Drug: doxorubicin; Drug: epirubicin; Drug: pirarubicin; Drug: cyclophosphamide; Drug: albumin-bound paclitaxel
- AC followed by taxanes (Active Comparator): A (doxorubicin, epirubicin or pirarubicin) and C (cyclophosphamide) for 4 cycles followed by paclitaxel or docetaxel for 4 cycles.
  Interventions: Drug: doxorubicin; Drug: epirubicin; Drug: pirarubicin; Drug: cyclophosphamide; Drug: paclitaxel; Drug: docetaxel

INTERVENTIONS:
Drug: doxorubicin — doxorubicin 50~60mg/m2, i.v., d1, q3w or q2w.
Drug: epirubicin — epirubicin 80~100mg/m2, i.v., d1, q3w or q2w.
Drug: pirarubicin — pirarubicin 40~50mg/m2, i.v., d1, q3w or q2w.
Drug: cyclophosphamide — cyclophosphamide 600mg/m2, i.v., d1, q3w or q2w.
Drug: albumin-bound paclitaxel — albumin-bound paclitaxel 260mg/m2, i.v., d1, q3w; 260mg/m2, i.v., d1, q2w; or 125mg/m2, i.v., d1, qw.
  Arms: AC followed by albumin-bound paclitaxel
Drug: paclitaxel — paclitaxel 175mg/m2, i.v., d1, q3w; 175mg/m2, i.v., d1, q2w; or 80mg/m2, i.v., d1, qw.
  Arms: AC followed by taxanes
Drug: docetaxel — docetaxel 80~100mg/m2, i.v., d1, q3w.
  Arms: AC followed by taxanes

SUMMARY:
This is a prospective, multi-center, real-world study designed to evaluate the efficacy and safety of albumin-bound paclitaxel versus paclitaxel or docetaxel in adjuvant treatment of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged from 18 to 70 years old;
2. Histologically confirmed as invasive breast cancer;
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
4. Participants achieved complete tumor resection by radical mastectomy, modified radical mastectomy or breast-conserving surgery with negative margins;
5. AC-T adjuvant chemotherapy is planned after breast cancer surgery;
6. Participants with HER-2 negative breast cancer at high risk of recurrence who meet any of the following conditions: 1) HR positive, and ≥4 positive lymph nodes or 1-3 positive lymph nodes with other risk of recurrence [such as high Ki67 expression (≥20%), T > 2 cm, age < 35 years, lymphovascular invasion, grade 3 histology]; 2) HR negative with positive lymph node or T > 2 cm;
7. LVEF ≥ 50%;
8. Participants had good compliance with the planned treatment and follow-up, understood the study procedures of this study, and signed informed consent form.

Exclusion Criteria:

1. In the past and present, participants with severe cardiac disease or discomfort , including but not limited: 1) High-risk uncontrolled arrhythmia, atrial tachycardia (heart rate > 100/min in resting state), significant ventricular arrhythmia (ventricular arrhythmia) or higher atrioventricular block (second-degree type 2 [Mobitz 2] atrioventricular block or third-degree atrioventricular block); 2) Angina pectoris requiring anti-angina medication; 3) Clinically significant valvular heart disease; 4) ECG showing transmural myocardial infarction; 5) Uncontrolled hypertension (eg systolic blood pressure > 180mm Hg or diastolic blood pressure > 100mmHg); 6) Myocardial infarction; 7) Congestive heart failure;
2. Participants who have received prior any systematic treatment for breast cancer;
3. Participants with bilateral invasive breast cancer;
4. Breast cancer with distant metastasis;
5. Grade 2 or higher Sensory or motor neurotoxicity was present as assessed by CTCAE V5.0;
6. Participants have the following serious illnesses or medical conditions, including but not limited: 1) History of serious neurological or psychiatric disorders, including psychosis, dementia, or epilepsy, that prevent understanding and informed consent; 2) Active uncontrolled infection; 3) Active peptic ulcer, unstable diabetes;
7. Previous or current existence of other malignant tumors other than breast cancer;
8. Severe liver and kidney dysfunction;
9. The presence of any myelodysplastic and other hematopoietic disorders;
10. Participants who are known to be allergic to the active or other components of the study treatment;
11. Participants who are pregnant, breastfeeding, or refuse to use adequate contraception prior to study entry and for the duration of study participation;
12. Participants who were judged by the investigator to be unsuitable for this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
5-year invasive disease-free survival (IDFS) rate | up to 60 months
  Invasive disease free survival was defined as the time from enrollment until the date of first occurrence of one of the following events: invasive ipsilateral breast tumor recurrence, local/regional invasive recurrence, distant recurrence (including first metastasis), invasive contralateral breast cancer, second primary invasive cancer (nonbreast, not including squamous or basal cell skin cancers, or new in situ carcinomas of any site), or death from any cause. 5-year IDFS rate is thepercentage of participants with IDFS from enrollment through 5 years.

SECONDARY OUTCOMES:
IDFS | up to 60 months
  Invasive disease free survival was defined as the time from enrollment until the date of first occurrence of one of the following events: invasive ipsilateral breast tumor recurrence, local/regional invasive recurrence, distant recurrence (including first metastasis), invasive contralateral breast cancer, second primary invasive cancer (nonbreast, not including squamous or basal cell skin cancers, or new in situ carcinomas of any site), or death from any cause.
overall survival (OS) | up to 60 months
  OS was defined as the time from enrollment assignment to death as a result of any cause.
3-year invasive disease-free survival (IDFS) rate | up to 36 months
  3-year IDFS rate is the percentage of participants with IDFS from enrollment through 3 years.
Incidence and severity of adverse events | up to 60 months
  Adverse events as assessed by NCI-CTCAE V5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, ChineseAMS, Beijing, Beijing Municipality, China